CLINICAL TRIAL: NCT03735199
Title: 3D Printed Scaffold Device for Ridge Preservation After Tooth Extraction - A Randomised Controlled Clinical Trial
Brief Title: 3D Printed Scaffold Device for Ridge Preservation After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Dental Centre, Singapore (Other)
Collaborators: Osteopore International (Unknown)
Responsible Party: Principal Investigator, Goh Bee Tin, Senior Consultant, Department of Oral & Maxillofaical Surgery, Clinical Associate Professor, Director of Research, NDCS, National Dental Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTGCoD-2001
Record Dates: First submitted 2018-10-03; First posted 2018-11-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bone Resorption After Tooth Extraction
Keywords: 3D Printed Scaffold Device

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCL-TCP scaffold (Experimental): During the surgery, the PCL-TCP scaffold will be shaped by cutting and shaving with a scalpel so as to fit the extraction socket snugly at the crestal half to two-thirds aspect. A Geistlich Bio-Gide collagen membrane will be placed over the scaffold at the crestal aspect of the socket. The periosteum of the buccal flap will then be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.
  Interventions: Device: PCL-TCP scaffold; Device: Geistlich Bio-Gide collagen membrane
- Geistlich Bio-Gide collagen membrane (Active Comparator): No space filler will be inserted in the extraction socket but similar to the test group, a Geistlich Bio-Gide collagen membrane will be placed over the crestal aspect of the socket and the periosteum of the buccal flap will be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.
  denture overlying the extraction site will be completely relieved.
  Interventions: Device: Geistlich Bio-Gide collagen membrane

INTERVENTIONS:
Device: PCL-TCP scaffold — During the surgery, the scaffold will be shaped by cutting and shaving with a scalpel so as to fit the extraction socket snugly at the crestal half to two-thirds aspect. A collagen membrane will be placed over the scaffold at the crestal aspect of the socket. The periosteum of the buccal flap will then be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.
  Arms: PCL-TCP scaffold
Device: Geistlich Bio-Gide collagen membrane — A collagen membrane will be placed over the crestal aspect of the socket and the periosteum of the buccal flap will be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.

SUMMARY:
Following tooth extraction, the socket heals naturally with bone in 1 to 2 months. This healing process occurs with substantial reduction of the original height and width of the alveolar ridge. In a significantly resorbed ridge, bone augmentation procedures are necessary before dental implant placement. Autogenous bone is the gold standard for this purpose but the harvesting procedure results in additional morbidities and expenses. Ridge preservation techniques have been introduced, using xenografts, allografts or synthetic materials to fill the tooth socket immediately after extraction. While the current materials used have improved ridge dimensions to various extents, their osteoconductivity is suboptimal and unpredictable. They do not reduce vertical resorption of the bony walls and often interfered with the normal healing process. Polycaprolactone - tricalcium phosphate (PCL-TCP) is a bioactive, bioresorbable composite polymer that is non-toxic and tissue-compatible. This study will test the use of a novel 3D printed PCL-TCP device for ridge preservation, leveraging on its 3D shape that fits snugly in the tooth socket, high porosity and bioactivity to promote osteogenesis and reduce resorption. The hypothesis is that the insertion of a PCL-TCP scaffold in extraction sockets allows normal bone healing and better maintenance of ridge dimensions after 6 months compared to extraction sockets without a space filler. This will be a prospective, randomized controlled clinical trial in patients who require single tooth extraction and replacement with a dental implant. The study will compare the ridge dimensions and the quality and quantity of bone formed in tooth sockets, using histology and microcomputed tomography, in both groups after 6 months. The PCL-TCP scaffold to be used in this study will be fabricated by a local spin-off company, Osteopore International Pte Ltd. The market potential for this device is tremendous due to a growing demand for tooth replacement from an ageing population worldwide.

DETAILED DESCRIPTION:
This will be a prospective, non-blinded randomized controlled clinical trial in adult patients who require single tooth extraction and who are suitable for dental implant therapy after extraction. The participants will be randomised by a clinician, using sealed envelopes that has been prepared by an independent party, to either the test or control group on a 1:1 ratio:

Test Group: insertion of PCL-TCP scaffold after tooth extraction Control Group: no space filler after tooth extraction

Proposed study interventions 110 patients who give written consent to participating in the study will be recruited from the Departments of Oral & Maxillofacial Surgery and Restorative Dentistry at the NDCS.

Patient may re-participate in the study for a different suitable teeth site. The re-participation(s) may take place on the same or a separate visit.

Pre-extraction Preparation Dental models and standardised dental radiographs, including periapical and orthopantomogram, will be taken. A customised acrylic dental stent will be fabricated as a reference tool for standardised measurement of ridge dimensions. Three markings will be made (mesio-buccal, mid-buccal, disto-buccal) on the acrylic stent at the intended extraction site.

Surgical Extraction and Socket Management

Under local anesthesia, a trapezoidal buccal mucoperiosteal flap will be raised and an atraumatic extraction of the tooth will be performed. The tooth socket will be thoroughly debrided and any granulation tissue will be curetted out. The acrylic measuring stent will then be positioned by fitting it to the adjacent teeth and the following measurements will be taken using a periodontal probe (PCPUNC15; Hu-Friedy USA):

Ridge height This will be measured indirectly as the vertical distance from each reference marking on the stent to the marginal bone of the tooth socket at the mesio-buccal, mid-buccal and disto-buccal aspects (Figure 1) and will recorded as RHmeb1, RHmib1 and RHdb1 respectively.

Ridge width This will be the horizontal distance from the buccal aspect to the lingual/ palatal aspect of the alveolar crest at the mid-buccal region of the extraction socket (RW1).

All measurements will be taken by 2 independent parties. Measurements that differ by less than or equal to 1mm will be averaged. Those that differ by more than 1mm will be repeated and a consensus will be reached by the parties. All measurements will be approximated to the nearest 0.5 mm.

The extraction sockets will be managed differently for the test and control groups:

Test Group

PCL-TCP scaffold:

The PCL-TCP scaffolds will be supplied by Osteopore International (Singapore). The scaffolds will be fabricated by the latest FDM techniques (FDM 3000; Stratasys, Eden Prairie, MN), in a class 10K clean room environment. Each scaffold will have a lay-down pattern of 0°/60°/120°, porosity of 70% and will be conical in shape. The scaffolds will a typical honeycomb structure with interconnected equilateral triangles of regular porous morphology. They will be individually packed and sterilized using gamma irradiation.

One or more suitable size scaffold(s) will be chosen (small or large) based on the tooth to be extracted. During the surgery, the scaffold will be shaped by cutting and shaving with a scalpel so as to fit the extraction socket snugly at the crestal half to two-thirds aspect. A collagen membrane will be placed over the scaffold(s) at the crestal aspect of the socket. The periosteum of the buccal flap will then be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.

Control Group No space filler will be inserted in the extraction socket but similar to the test group, a collagen membrane will be placed over the crestal aspect of the socket and the periosteum of the buccal flap will be incised to allow a tension-free primary closure with 4/0 Vicryl® suture.

A periapical radiograph of the extraction site will be taken using standardised settings immediately postoperatively. A 5-day course of Amoxicillin (or Clindamycin if the patient is allergic to Penicillin) will be prescribed together with an analgesic and chlorhexidine digluconate 0.2% mouthrinse. The sutures will be removed 1 week postoperatively. The surgical site will be examined clinically for any signs of infection or wound dehiscence. A temporary denture will be issued where necessary. The denture overlying the extraction site will be completely relieved.

Stage I Dental Implant Surgery Surgical placement of a dental implant will be performed at 6 months after tooth extraction. Radiographs, including a periapical of the study site, will be taken before the surgery. Following local anaesthesia and elevation of a full-thickness mucoperiosteal flap, the site will be clinically observed for any signs of inflammation, infection and presence of fibrous or bone tissue ingrowth. The same customised acrylic stent used for the case at the time of the tooth extraction will be used for measuring new ridge height dimensions in a manner similar to that described previously. Readings will be recorded as RHmeb2, RHmib2 and RHdb2. Ridge width will be measured as previously described and recorded as RW2.

The patient in either the test or control group will be taken out of the study at this stage if it is found that the extraction site has undergone extensive bone resorption such as to warrant simultaneous bone grafting with implant placement or pre-implant bone grafting with delayed implant placement.

Prior to implant placement, a core of bone of 2 mm diameter and 6 mm length at the healed extraction site will be obtained using a trephine bur (3i Implant Innovations Inc.; USA). The core of bone will be fixed and stored in 10% neutral buffered formalin and sent for microcomputed tomography (micro CT) scanning and histological preparation.

The implant site will be prepared using successive drills, according to the Straumann® (Institut Straumann AG, Basel, Switzerland) dental implant surgical protocol. A dental implant (Straumann® Bone Level) of the appropriate length and diameter will then be inserted at an insertion torque of between 20 Ncm and 40 Ncm. After placement of the dental implant, Implant Stability Quotient (ISQ) will be measured by Resonance Frequency Analysis (RFA) using the Osstell® machine. A cover screw will be placed over the implant. A releasing incision of the periosteum will be done if necessary and the surgical wound will be closed primarily with 4/0 Vicryl®.

A 5-day course of Amoxicillin (or Clindamycin if the patient was allergic to Penicillin) will be prescribed postoperatively, together with an analgesic and chlorhexidine digluconate 0.2% mouthrinse. The sutures will be removed 1 week postoperatively. The surgical site will be examined clinically for any signs of infection or wound dehiscence. The denture overlying the extraction site will be completely relieved.

Stage II Dental Implant Surgery This will be performed 3 months after Stage I dental implant surgery. The site will be observed for any signs of inflammation, infection as well as clinical stability of the dental implant. ISQ will be measured by RFA using the Osstell® machine before attachment of the healing abutment.

Analyses

1. Clinical Analysis of Bone Resorption

   The amount of vertical bone resorption in millimeters (mm) at 3 aspects will be calculated:

   Mesio-buccal: RHmeb2 - RHmeb1 Mid-buccal: RHmib2 - RHmib1 Disto-buccal: RHdb2 - RHdb1

   The amount of horizontal bone resorption in millimeters at the mid-buccal aspect will be calculated:

   RW1 - RW2
2. ISQ ISQ at Stage I and II dental implant surgery will be measured by 2 independent parties using RFA for both the test and control groups.
3. Radiopacity Grading Scale The degree of radiopacity of the tooth socket observed on the periapical radiograph taken at 6 months post-extraction in both the test and control groups will be graded according to the following scale.

1 = radiolucent similar to tooth socket* 2 = increased radiopacity but less than surrounding bone 3 = increased radiopacity similar to surrounding bone 4 = increased radiopacity more than surrounding bone

* compared with baseline periapical taken of tooth socket immediately after surgical extraction

The investigator performing the grading will be blinded to the grouping of the radiographs.

4) Micro CT Analysis

Quantitative analysis of bone regeneration in the test and control specimens will be performed using micro CT (SkyScan 1076, Kontich, Belgium). The specimens, consisting of 2 mm diameter by 6 mm length core of bone, will be placed in a sample holder and scanned through 180° at a spatial resolution of 30μm. The image data from the scanned planes will be subsequently thresholded, reconstructed to create 3D images and analysed using VGStudio Max 1.1 and CT Analyzer software (Volume Graphics GmbH, Heidelberg, Germany). The region of interest (ROI) will be defined by the boundaries of the specimen of each slice. The ROI will be interpolated through the entire length of the specimen to form the volume of interest (VOI). To select the area for bone, a bone-defining threshold will be set manually and kept constant for all the images. The percentage bone volume (BV%) will be obtained from the ratio of bone volume (BV) to total volume (TV):

BV% = BV/ TV

5) Histological Analysis After micro CT scanning, the specimens will be dehydrated in a graded series of ethanol, embedded in glycol methacrylate resin and polymerised. The block will be trimmed to remove excess plastic with an industrial vertical band saw and cut along its long axis with a diamond band saw (EXAKT standard saw). Ground polished sections of 10 μm thickness will be made using the EXAKT micro grinder system (EXAKT Technologies, Inc., Oklahoma City, OK) and will be subsequently stained with Hematoxylin and Eosin (H&E), Goldner's trichrome and von Kossa for descriptive histology.

(iii) Methods for protecting against other sources of bias (eg. blinding or masking. If blinding is not possible, please explain why and give details of alternative methods proposed or implications for interpretation of trials results)

As this study will compare the use of a device in a tooth socket (test group) versus no device (control group), blinding is not possible. To reduce bias, 2 independent parties will perform the ridge dimension and ISQ measurements.

The investigator performing the Radiopacity Grading Scale will be blinded to the grouping of the radiographs. Blinding for the micro CT and histology analyses is not possible as the presence/ absence of PCL-TCP scaffold will be obvious in the specimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be above 21 and below 70 years of age (both inclusive)
* Patient must be of ASA I or ASA II classification
* Patient who requires single tooth extraction
* Patient whose tooth to be extracted is bounded by adjacent teeth
* Patient who is suitable for dental implant therapy after extraction
* Patient with any pre-existing infection or abscess at the site of tooth extraction must be treated and resolved first prior to inclusion in the study

Exclusion Criteria:

* Patient with known allergy to biopolymer materials
* Patient who are smokers
* Patient who has undergone therapeutic radiation for head and neck malignant disease
* Maxillary lateral incisor and molars; or mandibular central and lateral incisor extraction sites
* Extraction sites with insufficient vertical bone height for implant placement without additional bone grafting (such as sinus lift procedure)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge resorption | 6 months post-extraction
  This will be measured indirectly as the vertical distance from each reference marking on the stent to the marginal bone of the tooth socket at the mesio-buccal, mid-buccal and disto-buccal aspects

SECONDARY OUTCOMES:
Quality of bone tissue formed in tooth sockets | 6 months post-extraction
  Descriptive histology will be performed for the test and control groups after 6 months.
Quantity of bone tissue formed in tooth sockets | 6 months post-extraction
  Micro-CT scans will be performed for the test and control groups after 6 months. Bone Volume % will be calculated.
Stability of dental implant | 6 months post-extraction
  Implant Stability Quotient (ISQ) will be measured by Resonance Frequency Analysis (RFA) using the Osstell® machine.
Healing and inflammatory response in tooth sockets | 6 months post-extraction
  via clinical observation and histology

CONTACTS AND LOCATIONS:
Overall Officials: Bee Tin Goh, Principal Investigator — National Dental Centre, Singapore
Locations (1):
- National Dental Centre Singapore, Singapore, Singapore

DOCUMENTS (1):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03735199/Prot_000.pdf